CLINICAL TRIAL: NCT01502839
Title: Differentiating Between Mild Traumatic Brain Injury And Behavioral Health Conditions: The Role of The Neurobehavioral Symptom Inventory
Brief Title: Role of NSI in Differentiating Between Mild Traumatic Brain Injury And Behavioral Health Conditions
Status: Terminated | Type: Observational
Why Stopped: Unable to complete the data collection for this study.
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 11-0219
Record Dates: First submitted 2011-12-09; First posted 2012-01-02 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2012-12

CONDITIONS: Traumatic Brain Injury; Post-Concussive Symptoms; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OEF/OIF Veterans: Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) Veterans
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This retrospective data analysis will rely on data obtained from chart review.

SUMMARY:
The purpose of this study is to examine differences in post-concussive (PC) symptom endorsement among four groups of Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) Veterans: those with a history of target, service-related, mild traumatic brain injury (mTBI) and co-occurring posttraumatic stress disorder (PTSD) (Group 1); those with a history of target, service-related, mTBI only (Group 2); those with PTSD only (Group 3); and those with no history of target, service-related, mTBI or PTSD (Group 4) by examining scores on the Neurobehavioral Symptom Inventory (NSI). Support for this study is provided by previous research highlighting the complex relationship between mTBI, PTSD and subsequent PC symptom endorsement (Brenner et al. 2010; Terrio et al, 2009).

HYPOTHESES ARE AS FOLLOWS:

1. Individuals with a history of target, service-related, mTBI only (Group 2) and individuals with PTSD only (Group 3) each will report significantly more PC symptoms, as measured by NSI total scores, when compared to those with no history of service-related mTBI or PTSD (Group 4).
2. Individuals with co-occurring target, service-related, mTBI history and PTSD (Group 1) will report significantly more PC symptoms, as measured by total NSI scores, than either those with target, service-related, mTBI only (Group 2) or those with PTSD only (Group 3).

DETAILED DESCRIPTION:
Archival data will be collected from all OEF/OIF Veterans who were seen in the VA ECHCS TBI Clinic by Nancy Cutter, M.D. and her team between January 1, 2009 and December 31, 2010. Electronic Medical Record (EMR) progress note titles "OEF/OIF TBI 2nd Level Evaluation Consult Report" and "TBI Consult Report" will be used to identify potential subjects.

Power is based on the primary hypothesis that those with PTSD only (Group 3) and those with target, service-related mTBI only (Group 2) will have significantly more PC symptom reporting than those with no history of target, service-related mTBI or PTSD (Group 4). Belanger et al. (2010) reported a standard deviation of 15.3 on the NSI total score in a sample of 134 mTBI subjects. Assuming variability similar to the Belanger study, a significance level of 0.025 to correct for the two comparisons and 80% power, 180 subjects per group will detect a clinically significant difference of 5 points. For simplicity, this was calculated using a two-sided, two-sample t-test. Given that we are modeling all four groups together, pooled standard error estimates will be used, which will result in slightly higher power.

All analyses will assume a two-sided test of hypothesis with an overall significance level of 0.05, unless otherwise noted, and will be performed in either Statistical Analysis Software (SAS) v9.2 or above (SAS Institute, Inc., Cary, NC).

Demographic characteristics will be reported as means and standard deviations; medians and ranges; and proportions, as appropriate. Likewise, characteristics will be compared between the four aforementioned subject groups using Analysis of Variance (ANOVA), chi-square tests and/or nonparametric tests as appropriate.

Hypothesis 1: An ANOVA with reference cell coding will be utilized to model NSI total score as a function of the four groups (Group 1: Individuals with co-occurring target, service-related, mTBI and PTSD; Group 2: those with target, service-related, mTBI only; Group 3: those with PTSD only; and Group 4: those with no history of target, service-related, mTBI or PTSD). Potential confounders will then be assessed individually by adding them to the model with the groups. If any of the group parameter estimates changes by more than 10% with the inclusion of the potential confounder, the variable will be utilized in the final model. Once the final model is determined, a contrast will be set up within the model to test (1) PTSD only vs. Neither and (2) target, service-related, mTBI only vs. Neither, a Bonferroni correction will be employed such that the significance level will be adjusted to 0.025 for these two primary tests. Estimated mean differences will be reported with 95% CIs. Potential confounding variables to be considered are: age; gender; total number of deployments; time since last deployment; time since earliest documented mTBI; time since target, service-related, mTBI; and total number of mTBIs.

Hypothesis 2: Within the same final model above, a contrast will be used to test (1) those with co-occurring target, service-related, mTBI and PTSD vs. PTSD only and (2) those with co-occurring target, service-related, mTBI and PTSD vs. target, service-related, mTBI only.

ELIGIBILITY:
Inclusion criteria for all groups includes:

* Veteran must be between the ages of 18 to 60
* Veteran must have at least one OEF/OIF deployment
* Veteran must have received an OEF/OIF TBI 2nd Level Evaluation though the VA ECHCS TBI Clinic

Specific inclusion/exclusion criteria for each group are as follows:

Inclusion Criteria:

Group 1: (Both) Co-Occurring PTSD and target, service-related, mTBI

PTSD:

* Clinician confirmed PTSD diagnosis and continuous documentation of symptoms related to PTSD diagnosis within 1 year prior to being seen in the TBI Clinic, or
* Clinician confirmed PTSD diagnosis within 1 year prior to being seen in the TBI Clinic, or
* Clinician confirmed PTSD diagnosis within 60 days after being seen in TBI Clinic
* Target, service-related, mTBI
* Veterans with clinician confirmed target, service-related, mTBI per OEF/OIF TBI 2nd Level Evaluation Consult Report note in EMR

Group 2: (mTBI only) History of target, service-related, mTBI but with no diagnosis of PTSD

* PTSD:
* Veterans with no history of clinician confirmed PTSD diagnosis, or
* Veterans with previous clinician confirmed PTSD diagnosis , but without continuous documentation of PTSD symptoms within 1 year prior to being seen in the TBI clinic
* Target, service-related, mTBI
* Veterans with clinician confirmed target, service-related, mTBI per OEF/OIF TBI 2nd Level Evaluation Consult Report note in EMR

Group 3: (PTSD only) No history of target, service-related, mTBI but with a diagnosis of PTSD

* PTSD:
* Clinician confirmed PTSD diagnosis and continuous documentation of symptoms related to PTSD diagnosis within 1 year prior to being seen in the TBI Clinic, or
* Clinician confirmed PTSD diagnosis within 1 year prior to being seen in the TBI Clinic, or
* Clinician confirmed PTSD diagnosis within 60 days of being seen in TBI Clinic
* TBI:
* Veterans with no history of clinician confirmed diagnosis of target, service-related, mTBI
* Veterans with clinician confirmed mTBI prior to service and without continuous documentation of related symptoms within 1 year of being seen in the TBI Clinic

Group 4: (Neither) No history of target, service-related, mTBI and no diagnosis of PTSD

* PTSD:
* Veterans with no history of clinician confirmed PTSD diagnosis, or
* Veterans with previous clinician confirmed PTSD diagnosis , but without continuous documentation of PTSD symptoms within 1 year of being seen in the TBI clinic
* TBI:
* Veterans with no clinician confirmed diagnosis of target, service-related, mTBI

Exclusion Criteria:

* Those not meeting inclusion criteria as listed above, and
* Veterans with any history of clinician confirmed moderate or severe TBI, and
* Veterans with no NSI in TBI Consult Report note in EMR
* Veterans with documentation of any neurological event or disorder other than mTBI
* Veterans with positive brain imaging

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Archival data will be collected from all OEF/OIF Veterans who were seen in the VA ECHCS TBI Clinic by Nancy Cutter, M.D. and her team between January 1, 2009 and December 31, 2010. Electronic Medical Record (EMR) progress note titles "OEF/OIF TBI 2nd Level Evaluation Consult Report" and "TBI Consult Report" will be used to identify potential subjects.
Sampling Method: Non-Probability Sample
Enrollment: 887 (Actual)
Dates: Start 2011-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Inventory | 1 day (NSI was administered 1 time during clinical visit and documented in EMR as described below)
  The Neurobehavioral Symptom Inventory (NSI; Cicerone & Kalmar, 1995)is a 22-item self-report measure of PC symptoms recommended for use among military personnel by the Department of Defense (DoD). Subject responses to all 22 items will be extracted from each subject's TBI Consult Report note provided in her/his Electronic Medical Record (EMR).
  Estimated time to collect all data from this retrospective chart review is 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Signoracci, Ph.D., Principal Investigator — VA Eastern Colorado Health Care System
Locations (1):
- VA Eastern Colorado Health Care System, Denver, Colorado, United States